CLINICAL TRIAL: NCT00425256
Title: Evaluate the Safety and Efficacy of Bremelanotide in Women With Female Sexual Arousal Disorder (FSAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Collaborators: King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Robert Jordan, Palatin Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PT-141-2005-53
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Sexual Arousal Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — bremelanotide

INTERVENTIONS:
Drug: Bremelanotide

SUMMARY:
This 8 week at home study is designed to explore efficacy endpoints and evaluate the safety of intranasal Bremelanotide in women with Female Sexual Arousal Disorder. Efficacy will be assessed vs. a parallel placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal and in general good health
* In a stable relationship with a male partner for at least 6 months
* Willing to attempt sexual activity once a week with your partner

Ages: 21 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Quality of Life Medical & Research Center, LLC, Tucson, Arizona
  - University of California, Department of Family and Preventative Medicine, La Jolla, California
  - Downtown Women's Health Care, Denver, Colorado
  - Coastal Connecticut Research, New London, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Clinical Study Center, Fort Myers, Florida
  - Center For Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Center for Sexual Medicine at Sheppard Pratt, Baltimore, Maryland
  - Advanced Biomedical Research, Inc, Hackensack, New Jersey
  - The Center for Female Sexuality, Purchase, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Medford Women's Clinic, LLP, Medford, Oregon
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Advanced Clinical Therapies, Inc., West Reading, Pennsylvania
  - Accelovance, Houston, Texas
  - Women's Clinical Research Center, Seattle, Washington